CLINICAL TRIAL: NCT02705495
Title: Segmental and Ear Acupuncture for Prevention of Recurrent Urinary Tract Infections(SARUTI Study): a Multicenter Randomized Controlled Trial
Brief Title: Acupuncture for Prevention of Recurrent Urinary Tract Infections.
Acronym: SARUTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SARUTI V1.6
Record Dates: First submitted 2016-02-01; First posted 2016-03-10 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Active Comparator): 12 acupuncture treatments according to a standardized protocol, plus recommendation for use of cranberry products
  Interventions: Other: acupuncture; Drug: Cranberry products
- Control (Other): Recommendation for use of cranberry products only
  Interventions: Drug: Cranberry products

INTERVENTIONS:
Other: acupuncture — Acupuncture will be performed according to the physiological concept of segmental acupuncture. A fixed schema of acupuncture points will be used irrespective of TCM diagnosis. Needles will be inserted approximately 10 mm under the skin. The "deqi sensation" (a sensation described as numbness, heaviness, and distension) may be obtained, but will not be specifically aimed for. The acupuncture protocol includes body and ear acupuncture.
  Arms: acupuncture
Drug: Cranberry products — Participants will receive Cranberry products (Urgenin Blasenkapseln® and/or Alpinamed Preiselbeer Granulat ®) - use is recommended but not obligatory.
  Other Names: Cranberry tablets and juice

SUMMARY:
In this multi-centre prospective randomized controlled trial the efficacy of segmental acupuncture in the prevention of recurrent urinary tract infections will be assessed. The study (acupuncture) group will receive 12 acupuncture treatments according to a standardized protocol, plus recommendation for use of cranberry products. The control group will receive recommendation for use of cranberry products only.

DETAILED DESCRIPTION:
1. Background 1.1. Urinary tract infection

   Urinary tract infections (UTI) are considered to be the most common bacterial infections, with approximately 80% of all UTIs occurring in women (1). Nearly one in three women is expected to have at least one episode of UTI by the age of 24 years and almost half of all women will experience one UTI during their lifetime (2). Recurrence affect approximately 20-30% of women with initial UTI, although recurrence rates vary widely (3).

   Recurrent UTIs are a common problem seen in clinical practice with important medical, social and financial implications. Prophylaxis of recurrent UTI is an ongoing challenge with several different management strategies being used (4). Low dose antibiotic prophylaxis for several months is effective, but fosters the development of antibiotic resistance of the causative microorganisms, but also the commensal flora.(4-8). In postmenopausal women vaginal estrogen therapy reduces symptomatic UTI episodes (1, 7). Further prevention strategies include the oral immunostimulant OM-89, the vaginal vaccine Urovac, lactobacilli prophylaxis, cranberry products and acupuncture (5, 7, 9).

   1.2.Cranberry products Cranberries have been used in the prevention of UTIs for many years. Cranberries contain two compounds with antiadherence properties that prevent fimbriated Escherichia coli from adhering to uroepithelial cells in the urinary tract (10). A recent review of 24 studies showed that the use of various cranberry products may have a small benefit for women with recurrent UTIs, although differences were not statistically significant (11).

   1.3. Acupuncture treatment The effectiveness of acupuncture has been established for a series of different conditions (12, 13). Up to date there are only two clinical trials studying the effect of acupuncture on the prevention of recurrent UTI, both conducted from the same research group. In one controlled trial of 67 adult women acupuncture was significantly more effective in preventing recurrent UTI compared to sham acupuncture than no treatment over an observation period of 6 months (14). In the second trial of 100 women acupuncture, administered twice weekly for 4 weeks, was significantly more effective in reducing the number of UTIs, but also in reducing the volume of residual urine. Acupuncture points were chosen according to patients´ individual diagnoses following traditional Chinese medical patterns. (15)
2. Study aims The present study aims to compare acupuncture treatment with standard treatment (recommendation for cranberry intake) in the treatment of uncomplicated recurrent UTIs in women and is designed as a prospective randomized controlled trial. We will assess the number of acute lower UTIs and subsequent treatment, the type and amount of self medication (cranberry products and others), health related quality of life and treatment satisfaction within a defined period of time.

   The results from this study will help to guide clinical practice with level I evidence and allow for effective treatment with regard to patient needs.
3. Methods/ Workplan This patient oriented non-profit clinical study is designed as a randomised controlled trial (6 months) with a follow-up period of 12 months.

Active recruitment: 12 months Randomised controlled trial: 6 months Short-term Follow-up: 12 months 3.1. Active recruitment After Ethics Committee approval patient recruitment will be started. Information material about the study, including contact details, will be provided at the outpatient clinics of the Dep. of Gynecology, the Dep. of Urology, and other local health care providers. During an initial visit patients will be informed about the study and inclusion and exclusion criteria will be evaluated. A structured medical history, including assessment of previous UTIs and other urogenital tract symptoms, will be obtained. After written informed consent is obtained participants will be randomized.

3.2. Randomized Controlled Trial (6 months)

At the time of randomization patients must not have signs or symptoms of an acute UTI, and must not currently receive antibiotic treatment. Randomizing will be done electronically (www.randomizer.at). Patients will be randomized in one of two treatment groups without stratification with a planned ratio of 1:1:

* Acupuncture treatment group 12 acupuncture treatments according to a standardized protocol plus recommendation for use of cranberry products
* Standard treatment group Recommendation for use of cranberry products only

Participants will be contacted bimonthly by telephone and asked about occurrence of UTIs, adverse events, study adherence and completion of study diary. At 6 months a control visit will be scheduled, the RCT will be completed and the main outcome parameter (number of women with no acute UTIs) and secondary outcome parameters (9.2.) will be assessed.

This will be followed by a 12 months short-term Follow-up. 3.3. Short-term Follow-up (12 months) Patients of both treatment groups may use any prophylactic treatment. Participants will be contacted bimonthly by telephone and asked about occurrence of UTIs, adverse events, and use of prophylactic and therapeutic treatments for UTIs.

The study is designed according to the 2010 CONSORT guidelines(16) and the STRICTA (Standards for Reporting Interventions in Clinical Trials of Acupuncture) guidelines (17).

ELIGIBILITY:
Inclusion Criteria:

* Recurrent UTIs: Two or more symptomatic UTIs within the last six 6 months or 3 or more infections within the last 12 months.
* At least two positive urine culture within this period of time
* No evidence of current UTI at the time of inclusion
* Women, Age 18 - 90 years
* Informed consent

Exclusion Criteria:

* Pregnancy
* Urogenital anatomical abnormality
* Evidence of kidney stones
* Indwelling catheter
* systemic diseases such as renal insufficiency, transplantation, diabetes, or immunodeficiency

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2015-05; Primary Completion 2021-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection (UTI) | 6 months
  Number of women with no acute UTI at 6 months

SECONDARY OUTCOMES:
Urinary symptoms | 6 months
  Occurrence of urinary symptoms without signs of UTI
Study diary | 6 months
  Use of cranberry products (type, length and amount) assessed by the study diary
Health related quality of life | 6 months
  Health related quality of life as measured by the Kings Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gerda Trutnovsky, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Gynecology/ Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No